CLINICAL TRIAL: NCT03304548
Title: Qualitative Research to Explore Patient Preference for Modes of Administration in Pulmonary Arterial Hypertension Treatments
Brief Title: Qualitative Research to Explore Treatment Preference in Pulmonary Arterial Hypertension (PAH) Subjects
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Adelphi Values (Unknown)
Responsible Party: Sponsor
Other Study IDs: 207754
Record Dates: First submitted 2017-10-02; First posted 2017-10-09 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Hypertension, Pulmonary
Keywords: Telephone interviews; Subcutaneous; Low-interventional; Qualitative research; PAH
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All subjects with PAH: A total of 8 to 10 US-English speaking PAH subjects will be recruited. They will take part in a 30-minute telephone concept elicitation interview. All interviews will be audio-recorded and transcribed verbatim.
  Interventions: Other: Telephone concept elicitation interview

INTERVENTIONS:
Other: Telephone concept elicitation interview — All interview questions are designed to be very open-ended in order to ascertain subjects' preferences in an un-biased manner (as possible), with additional probes only being used when necessary to ensure all concepts of interest are covered. Subjects will be asked a series of broad, open-ended questions designed to encourage them to talk openly and as spontaneously as possible about their experience of taking oral treatment(s) for their PAH.

SUMMARY:
GlaxoSmithKline (GSK) is embarking on a clinical program to assess the treatment of PAH with an Angiotensin converting enzyme 2 (ACE2). This new treatment may require subcutaneous administration, in comparison to current treatments which are taken orally. Hence, GSK would like to conduct this qualitative interview study with PAH subjects to explore subject's perspective and preferences for various modes of treatment administration (daily or weekly subcutaneous injection versus current treatment options). This will be a qualitative study comprising the conduct of semi-structured telephone concept elicitation interviews with 8 to 10 PAH subjects (each approximately 30 minutes in duration) in the United States (US).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age.
* Subject is willing and able to provide written informed consent.
* Subject must have a diagnosis of symptomatic Pulmonary Arterial Hypertension Type I as per the World Health Organization (WHO) clinical classification system.
* Subject must have the cognitive and linguistic capabilities sufficient to allow them to actively participate in an interview lasting 30 minutes.

Exclusion Criteria:

* Subject has a diagnosis of other cardiac or pulmonary disease.
* Subject has a Type II-V diagnosis of PAH, as per the WHO clinical classification system.
* Subject is currently receiving treatment for PAH via modes of administration other than intravenously or orally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample of 8 to 10 US-English speaking subjects will be recruited. Recruitment will be facilitated by a third-party vendor in the US. A purposive approach to sampling will be employed to ensure subjects with a range of demographic and clinical characteristics are recruited.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects who preferred subcutaneous injection versus current treatment options | Up to 30 minutes
  All recruited subjects will take part in a 30-minute telephone interview. Subjects will be given brief descriptions of hypothetical injection and inhaled treatments and will be asked for their thoughts towards these treatments individually.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Boston, Massachusetts, United States

REFERENCES:
- See also: Results for study 207754 can be found on the GSK Clinical Study Register. — https://www.gsk-studyregister.com/study/6028